CLINICAL TRIAL: NCT00942188
Title: Phase 2 Randomized, Double-blind, Placebo Controlled, Parallel Design Study in Patients With Type 2 Diabetes Mellitus Who Are Stable on Diet and Exercise, With or Without Metformin Monotherapy.
Brief Title: A Study of LY2189102 in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13286; H9C-MC-BBDK (Other: Eli Lilly and Company)
Record Dates: First submitted 2009-07-17; First posted 2009-07-20 (Estimated); Results first posted 2018-03-13 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — LY2189102

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 0.6 milligrams (mg) LY2189102 (Experimental)
  Interventions: Drug: LY2189102
- 18 mg LY2189102 (Experimental)
  Interventions: Drug: LY2189102
- 180 mg LY2189102 (Experimental)
  Interventions: Drug: LY2189102
- Placebo (Placebo Comparator): 0.9% Sodium Chloride
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY2189102 — Participants received 2 subcutaneous (SC) injections weekly for 12 weeks.
  Arms: 0.6 milligrams (mg) LY2189102; 18 mg LY2189102; 180 mg LY2189102
Drug: Placebo — Participants received 2 SC injections weekly for 12 weeks.
  Arms: Placebo

SUMMARY:
Study to evaluate the safety, tolerability and efficacy of LY2189102 in patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Have Type 2 Diabetes and confirmed by fasting C-peptide levels greater than or equal to 0.8 nanograms per milliliter [ng/ml]), with duration of more than 3 months.
* Body mass index between 25 and 40 kilograms per square meter (kg/m2).
* Stable on diet and exercise alone, with or without metformin monotherapy (stable regimen or dose for at least 8 weeks).
* Drug-naïve or previous anti-diabetic pharmacotherapy use is allowed (for the latter, patient must have stopped taking pharmacotherapy greater than 12 weeks prior to screening and only if deemed appropriate by the investigator).
* Angiotensin converting enzyme inhibitors, angiotensin II receptor blockers, thiazide diuretics or calcium channel blockers are permitted for the treatment of hypertension or proteinuria.
* Glycated hemoglobin level between 7% and 10%.
* Baseline High-sensitivity C-reactive protein greater than or equal to 2 milligrams per liter (mg/L)
* Females of childbearing potential (not surgically sterilized and between menarche and 1 year post-menopause) must test negative for pregnancy at the time of enrollment based on a pregnancy test. Furthermore, sexually active female and male participants must agree to use 2 reliable methods of birth control during the study and for 3 months following the last dose of study drug.
* Reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures.

Exclusion Criteria:

* Current use of anti-diabetic pharmacotherapy (except metformin, under conditions specified in Inclusion Criteria above).
* Current treatment with anti-inflammatory drugs, including corticosteroids and non-steroidal anti-inflammatory drugs (100 mg per day or less of aspirin allowed).
* Within 60 days of the initial dose of the study drug, have received treatment with a drug that has not received regulatory approval for any indication.
* Presence of autoantibodies to glutamic acid decarboxylase 65 or islet-cell autoantibody-2.
* Evidence of tuberculosis as documented by a specific assay, medical history, and chest x-ray. A specific assay, (for example, tuberculin testing) will be conducted unless it is medically inappropriate. Exceptions include patients with a history of a positive specific assay for TB who have been treated with isonicotinyl hydrazine (documented) for at least 6 months, or patients with a previous diagnosis of TB who have been appropriately treated and can provide documentation.
* Symptomatic herpes zoster within 3 months of randomization.
* Show evidence of hepatitis C and/or positive hepatitis B surface antigen.
* Show evidence of human immunodeficiency virus and/or positive test of antibodies to human immunodeficiency virus (HIV).
* Received live or attenuated vaccine(s) within the previous 3 months prior to randomization or will receive within 3 months from the end of study.
* Screening serum creatinine greater than 2.0 milligrams per deciliter (mg/dL).
* Serum aspartate aminotransferase or alanine aminotransaminase concentration greater than 2x the upper limit of normal.
* Known allergies to LY2189102 or excipients.
* Previously completed or withdrawn from this study or any other study investigating LY2189102.
* Have donated blood of greater than 500 mL within the preceding 30 days and intend to donate within 3 months from the end of study.
* Have had other recent or ongoing signs of infection (for example, fever, current treatment with antibiotics).
* Experienced a serious bacterial infection within 6 months of randomization.
* Have a serious medical illness including but not limited to any cardiovascular, hepatic, respiratory, hematological, endocrine, or neurological disease, or any clinically significant laboratory abnormality.
* Have had lymphoma, leukemia, or any non-breast malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease.
* Have had a previous reaction to other biologics that, in the opinion of the investigator, puts the patient at serious risk.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2009-06; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (18):
- United States (18):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mobile, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Anaheim, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chula Vista, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., La Mesa, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Walnut Creek, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Washington D.C., District of Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miami Gardens, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Boise, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baltimore, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dearborn, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Philadelphia, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Arlington, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Antonio, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tomball, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salt Lake City, Utah
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Bihorel S, Fiedler-Kelly J, Ludwig E, Sloan-Lancaster J, Raddad E. Population pharmacokinetic modeling of LY2189102 after multiple intravenous and subcutaneous administrations. AAPS J. 2014 Sep;16(5):1009-17. doi: 10.1208/s12248-014-9623-6. Epub 2014 Jun 11. PMID 24912797

RESULTS

PARTICIPANT FLOW:
Groups:
- 0.6 mg LY2189102: Participants received 2 subcutaneous (SC) injections weekly for 12 weeks.
- 18 mg LY2189102; 180 mg LY2189102: Participants received 2 SC injections weekly for 12 weeks.
- Placebo: Participants received 2 SC injections of 0.9% sodium chloride weekly for 12 weeks.
Period: Overall Study
Arm/Group | 0.6 mg LY2189102 | 18 mg LY2189102 | 180 mg LY2189102 | Placebo
Started | 26 | 26 | 27 | 27
Completed | 22 | 16 | 18 | 23
Not Completed | 4 | 10 | 9 | 4
Not completed — Adverse Event | 0 | 3 | 2 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 1 | 1 | 0 | 0
Not completed — Lost to Follow-up | 2 | 1 | 2 | 0
Not completed — Withdrawal by Subject | 1 | 3 | 4 | 2
Not completed — Physician Decision | 0 | 0 | 1 | 0
Not completed — Sponsor Decision | 0 | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.6 mg LY2189102 | 18 mg LY2189102 | 180 mg LY2189102 | Placebo | Total
Number analyzed (Participants) | 26 | 26 | 27 | 27 | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.9 (6.75) | 53.7 (10.74) | 51.3 (9.17) | 52.9 (9.41) | 52.7 (9.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 17 | 15 | 20 | 67
  Male | 11 | 9 | 12 | 7 | 39
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 6 | 12 | 10 | 10 | 38
  African | 3 | 6 | 3 | 3 | 15
  Hispanic | 15 | 7 | 13 | 14 | 49
  East Asian | 0 | 1 | 0 | 0 | 1
  Other | 2 | 0 | 1 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26 | 26 | 27 | 27 | 106
Percentage of Glycosylated Fraction of Hemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin] — HbA1c: Hemoglobin A1c, glycosylated fraction of hemoglobin A (%)
  percentage of glycosylated hemoglobin | 7.540 (0.5596) | 7.950 (0.7002) | 8.271 (0.9380) | 7.824 (0.6557) | 7.882 (0.7544)
Fasting Glucose [Mean (Standard Deviation); unit: millimoles per liter (mmol/L)] | 8.152 (1.8154) | 9.106 (2.2001) | 10.300 (2.1440) | 9.339 (1.7315) | 9.208 (2.0688)
Fasting Insulin [Mean (Standard Deviation); unit: microinternational units per milliliter] | 15.083 (12.0562) | 15.034 (6.9383) | 13.989 (14.4076) | 15.120 (12.5253) | 14.821 (11.7856)
High-sensitivity C-reactive Protein (hsCRP) [Mean (Standard Deviation); unit: milligrams per liter (mg/L)] | 6.214 (6.2179) | 6.024 (4.4956) | 7.183 (6.9691) | 6.093 (4.5289) | 6.373 (5.5685)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per square meter (kg/m^2)] | 33.0 (3.73) | 33.7 (3.72) | 33.1 (4.02) | 32.5 (4.62) | 33.1 (4.01)
Number of Participants on Diet and Exercise Only [Count of Participants; unit: Participants]
  Diet and Exercise Only - Yes | 5 | 3 | 4 | 7 | 19
  Diet and Exercise Only - No | 21 | 23 | 23 | 20 | 87
Number of Participants on Anti-diabetic Medications [Count of Participants; unit: Participants] — The number of participants on anti-diabetic medications does not equal the total number of participants because some participants reported taking more than 1 anti-diabetic medication.
  Participants
    Biguanides | 20 | 23 | 22 | 20 | 85
    Glucagon-like Peptide (GLP) Analogs and Agonists | 1 | 0 | 0 | 0 | 1
    DPP-4 Inhibitors | 0 | 0 | 4 | 0 | 4
    Enhancers of Insulin Effects | 0 | 1 | 0 | 0 | 1
    Sufonylureas | 8 | 7 | 5 | 6 | 26

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Glycosylated Hemoglobin (HbA1c) at 12 Weeks
Description: Change in HbA1c from baseline following 12 weeks of therapy (that is, HbA1c at week 12 minus HbA1c at baseline). The Least Squares (LS) Mean Value was based on an analysis of covariance (ANCOVA) model with treatment and site as class variables and baseline HbA1c as a continuous covariate.
Time Frame: Baseline, 12 weeks
Population: Compliant set. All randomized participants receiving at least 11 doses of study drug were analyzed according to the treatment subjects were assigned.
Measure: Least Squares Mean (Standard Error); unit: percentage of glycosylated hemoglobin
Arm/Group | 0.6 mg LY2189102 | 18 mg LY2189102 | 180 mg LY2189102 | Placebo
Number analyzed (Participants) | 21 | 16 | 19 | 23
percentage of glycosylated hemoglobin | -0.457 (0.1454) | -0.561 (0.1530) | -0.428 (0.1379) | -0.183 (0.1315)

2. Secondary Outcome: Change From Baseline in Fasting Glucose at 12 Weeks
Description: Change in fasting glucose following 12 weeks of therapy (that is, fasting glucose at week 12 minus fasting glucose at baseline). The Least Squares (LS) Mean Value was based on an analysis of covariance (ANCOVA) model with treatment and site as class variables and baseline value as a continuous covariate.
Time Frame: Baseline, 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: millimole per liter (mmol/L)
Arm/Group | 0.6 mg LY2189102 | 18 mg LY2189102 | 180 mg LY2189102 | Placebo
Number analyzed (Participants) | 20 | 15 | 19 | 23
millimole per liter (mmol/L) | -0.873 (0.4802) | -1.270 (0.5299) | -0.629 (0.4591) | -0.019 (0.4404)
Statistical Analysis 1: Comparison: 0.6 mg LY2189102 vs Placebo; Test type: Superiority or Other; ANCOVA; LS Mean Difference = -0.854, 95% CI 2-sided [-1.94 to 0.23]
Statistical Analysis 2: Comparison: 18 mg LY2189102 vs Placebo; Test type: Superiority or Other; ANCOVA; LS Mean Difference = -1.252, 95% CI 2-sided [-2.48 to -0.03]
Statistical Analysis 3: Comparison: 180 mg LY2189102 vs Placebo; Test type: Superiority or Other; ANCOVA; LS Mean Difference = -0.610, 95% CI 2-sided [-1.76 to 0.54]

3. Secondary Outcome: Change From Baseline in Insulin Sensitivity (Fasting Insulin) at 12 Weeks
Description: Change in serum fasting insulin from baseline to endpoint (that is, serum insulin at week 12 minus serum insulin at week 0). The Least Squares (LS) Mean Value was based on an analysis of covariance (ANCOVA) model with treatment and site as class variables and baseline value as a continuous covariate.
Time Frame: Baseline, 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: microinternational Units per liter
Arm/Group | 0.6 mg LY2189102 | 18 mg LY2189102 | 180 mg LY2189102 | Placebo
Number analyzed (Participants) | 20 | 15 | 19 | 21
microinternational Units per liter | -1.589 (2.9549) | -0.918 (3.3206) | -0.229 (2.7836) | 1.405 (2.8722)
Statistical Analysis 1: Comparison: 0.6 mg LY2189102 vs Placebo; Test type: Superiority or Other; ANCOVA; LS Mean Difference = -2.995, 95% CI 2-sided [-9.82 to 3.83]
Statistical Analysis 2: Comparison: 18 mg LY2189102 vs Placebo; Test type: Superiority or Other; ANCOVA; LS Mean Difference = -2.324, 95% CI 2-sided [-10.21 to 5.56]
Statistical Analysis 3: Comparison: 180 mg LY2189102 vs Placebo; Test type: Superiority or Other; ANCOVA; LS Mean Difference = -1.635, 95% CI 2-sided [-9.16 to 5.89]

4. Secondary Outcome: Number of Participants With a Change From Baseline in Beta-Cell Function Measured by Glucose and Insulin Changes With the Mixed Meal Tolerance Test (MMTT) at 12 Weeks
Description: The number of participants with a change from baseline in glucose and insulin at 2 hours after the MMTT was analyzed. The MMTT measures glucose and insulin before and after a standardized meal is eaten. Glucose and insulin levels were measured before the MMTT and 2 hours after the MMTT.
Time Frame: Baseline, 12 weeks
Population: Full analysis set. All randomized participants who received at least 1 dose of the study drug according to the treatment they were assigned and for whom the data are considered sufficient and interpretable. Differences in Ns are due to either dropouts and no post-baseline measure or something occurred to the sample (for example, not taken, broke).
Measure: Number; unit: participants
Arm/Group | 0.6 mg LY2189102 | 18 mg LY2189102 | 180 mg LY2189102 | Placebo
Number analyzed (Participants) | 22 | 17 | 18 | 24
participants
  Glucose at 2 hours | 22 | 17 | 18 | 24
  Insulin at 2 hours | 22 | 17 | 18 | 24

5. Secondary Outcome: Change From Baseline in the Glycosylated Hemoglobin (HbA1c) at Week 10 and Week 12
Description: The change from baseline in HbA1c at week 10 (that is HbA1c at week 10 minus HbA1c at baseline) and week 12 (that is, HbA1c at week 12 minus HbA1c at baseline). The Least Squares (LS) Mean Value was based on an analysis of covariance (ANCOVA) model with treatment and site as class variables and baseline value as a continuous covariate.
Time Frame: Baseline, week 10, week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage glycosylated hemoglobin
Arm/Group | 0.6 mg LY2189102 | 18 mg LY2189102 | 180 mg LY2189102 | Placebo
Number analyzed (Participants) | 21 | 16 | 19 | 23
percentage glycosylated hemoglobin
  HbA1c at Week 10 | -0.456 (0.1459) | -0.555 (0.1541) | -0.413 (0.1412) | -0.186 (0.1322)
  HbA1c at Week 12: number analyzed (Participants) | 20 | 15 | 19 | 23
  HbA1c at Week 12 | -0.459 (0.1560) | -0.588 (0.1712) | -0.413 (0.1455) | -0.192 (0.1410)
Statistical Analysis 1: Comparison: 0.6 mg LY2189102 vs Placebo; Test type: Superiority or Other; ANCOVA — This is the estimated value for week 10 HbA1c; LS Mean Difference = -0.270, 95% CI 2-sided [-0.59 to 0.05]
Statistical Analysis 2: Comparison: 18 mg LY2189102 vs Placebo; Test type: Superiority or Other; ANCOVA — This is the estimated value for HbA1c at Week 10; LS Mean Difference = -0.369, 95% CI 2-sided [-0.74 to 0.00]
Statistical Analysis 3: Comparison: 180 mg LY2189102 vs Placebo; Test type: Superiority or Other; ANCOVA — This is the estimated value for HbA1c at Week 10; LS Mean Difference = -0.227, 95% CI 2-sided [-0.59 to 0.13]
Statistical Analysis 4: Comparison: 0.6 mg LY2189102 vs Placebo; Test type: Superiority or Other; ANCOVA — This is the estimated value for HbA1c at week 12; LS Mean Difference = -0.267, 95% CI 2-sided [-0.61 to 0.08]
Statistical Analysis 5: Comparison: 18 mg LY2189102 vs Placebo; Test type: Superiority or Other; ANCOVA — This is the estimated value for HbA1c at Week 12; LS Mean Difference = -0.396, 95% CI 2-sided [-0.79 to 0.00]
Statistical Analysis 6: Comparison: 180 mg LY2189102 vs Placebo; Test type: Superiority or Other; ANCOVA — This is the estimated value for HbA1c at week 12; LS Mean Difference = -0.221, 95% CI 2-sided [-0.59 to 0.15]

6. Secondary Outcome: Pharmacokinetics (PK) Maximum Serum Concentration (Cmax) of LY2189102 at End of Dosing (12 Weeks)
Description: The Cmax value measures the maximum serum concentration and is estimated for LY2189102. The values were generated as individual estimates from a population pharmacokinetics (PK) model.
  Placebo samples were not assayed for serum concentration of LY2189102 because the participants in the placebo treatment arm did not receive LY2189102 study drug.
Time Frame: Prior to and 1 and 3-4 days after the first dose, prior to every other dose, and 6 and 12 weeks after the last dose
Population: Full Analysis Set: All randomized participants who received at least 1 dose of the study drug according to the treatment they were assigned and for whom the data are considered sufficient and interpretable. Differences in Ns are due to either dropouts and no post-baseline measure or something occurred to the sample (for example, not taken, broke).
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | 0.6 mg LY2189102 | 18 mg LY2189102 | 180 mg LY2189102
Number analyzed (Participants) | 18 | 15 | 19
nanograms per milliliter (ng/mL) | 269.39 (88.23) | 6094.67 (2153.00) | 39994.74 (17880.45)

7. Secondary Outcome: PK: Area Under the Concentration Time Curve for Dosing Interval (Tau) at Steady State (AUCτ,SS) at End of Dosing (12 Weeks)
Description: Individual estimates of AUCtau at end of dosing generated from a population pharmacokinetic (PK) model.
Time Frame: Prior to and 1 and 3-4 days after the first dose, prior to every other dose, and 6 and 12 weeks after the last dose
Population: Compliant set. All randomized participants receiving at least 11 doses of study drug were analyzed according to the treatment subjects were assigned. Placebo samples were not assayed for serum concentration of LY2189102 because the participants in the placebo treatment arm did not receive LY2189102 study drug.
Measure: Mean (Standard Deviation); unit: nanogram*hour per milliliter (ng*h/mL)
Arm/Group | 0.6 mg LY2189102 | 18 mg LY2189102 | 180 mg LY2189102
Number analyzed (Participants) | 18 | 15 | 19
nanogram*hour per milliliter (ng*h/mL) | 45777.78 (14933.09) | 986533.33 (340965.83) | 6555789.47 (2934693.46)

8. Secondary Outcome: Pharmacokinetics Measured by Serum Concentration at End of Dosing (12 Weeks)
Description: Pharmacokinetics Measured by Serum Concentration at End of Dosing.
Time Frame: Prior to and 1 and 3-4 days after the first dose, prior to every other dose, and 6 and 12 weeks after the last dose
Population: All participants who received at least one dose of study drug and had evaluable PK data. Placebo samples were not assayed for serum concentration of LY2189102 because the participants in the placebo treatment arm did not receive LY2189102 study drug.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | 0.6 mg LY2189102 | 18 mg LY2189102 | 180 mg LY2189102
Number analyzed (Participants) | 18 | 15 | 19
nanograms per milliliter (ng/mL) | 252.83 (83.28) | 5532.00 (1991.28) | 35815.79 (15961.46)

ADVERSE EVENTS:
Arm/Group | 0.6 mg LY2189102 | 18 mg LY2189102 | 180 mg LY2189102 | Placebo
Serious Adverse Events (participants affected / at risk) | 1/26 | 1/26 | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 19/26 | 19/26 | 23/27 | 20/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.6 mg LY2189102 (N=26) | 18 mg LY2189102 (N=26) | 180 mg LY2189102 (N=27) | Placebo (N=27)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.6 mg LY2189102 (N=26) | 18 mg LY2189102 (N=26) | 180 mg LY2189102 (N=27) | Placebo (N=27)
Cardiac disorder (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Palpitations (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 3 (3) | 2 (2) | 3 (3)
Flatulence (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1) | 3 (3)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
Injection site haematoma (General disorders) | 0 (0) | 4 (4) | 0 (0) | 1 (1)
Injection site irritation (General disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (3)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Nasopharyngitis (Infections and infestations) | 5 (5) | 3 (3) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 3 (3) | 3 (4) | 1 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (2) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 4 (4) | 3 (3) | 2 (2)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 2 (2) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days